CLINICAL TRIAL: NCT00488072
Title: Preliminary Study to Explore the Effects of Mirtazapine on Appetite in Advanced Cancer Patients
Brief Title: Effects of Mirtazapine on Appetite in Advanced Cancer Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-0916; NCI-2011-02822 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-06-18; First posted 2007-06-19 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Advanced Cancer; Anorexia; Weight Loss; Insomnia
Keywords: Advanced Cancer; Anorexia; Weight Loss; Insomnia; Appetite; Mirtazapine; Placebo
MeSH Terms: conditions — Anorexia; Weight Loss; Sleep Initiation and Maintenance Disorders | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mirtazapine (Experimental): Mirtazapine 15 mg by mouth (PO) daily for 15 days; Day 22-29, increased to 30 mg PO daily.
  Interventions: Drug: Mirtazapine
- Placebo (Placebo Comparator): One placebo tablet by mouth daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirtazapine — 15 mg by mouth (PO) daily x 15 days; Day 22-29, increased to 30 mg PO daily.
  Arms: Mirtazapine
Drug: Placebo — One placebo tablet by mouth daily.
  Arms: Placebo

SUMMARY:
Primary objective: This is a preliminary study to determine if Mirtazapine in comparison to placebo will improve appetite in advanced cancer patients with anorexia and weight loss. An improvement of appetite is defined as a decrease of 2 in the appetite score from baseline on the Edmonton Symptom Assessment Scale (ESAS) at day 15 (+/-3 days).

Secondary objective-A: To determine if Mirtazapine in comparison to placebo will improve insomnia ( as measured by Pittsburgh Sleep Quality Index) on day 15 ( +/- 3 days), and day 29 ( +/- 3 days)

Secondary objective - B: To determine if Mirtazapine in comparison to placebo will improve other common symptoms such as pain, nausea and fatigue( as measured by ESAS), depression and anxiety ( as measured by Hospital Anxiety and Depression scale), and quality of life ( as measured by Functional Assessment of Anorexia/Cachexia Therapy ) in advanced cancer patients with anorexia/cachexia, on days 15 (+/-3 days), and 29 (+/-3 days)

Other Objectives:

To provide exploratory data on the effects of Mirtazapine on weight gain, and preservation/gain lean muscle mass ( anthropometric measurements and Bioelectric Impedance), on days 15 (+/-3 days), and 29 (+/-3 days).

To provide exploratory data on the effects of a Mirtazapine dose increase to 30 mg on decreased side effects of drug and increased appetite on day 29 (+/-3 days).

DETAILED DESCRIPTION:
Mirtazapine is a drug that is used to treat clinical depression. It is designed to cause hormones ("chemical messengers" such as norepinephrine and serotonin) to be released in the brain, while blocking certain molecules that cause nausea, nervousness, headache, insomnia, diarrhea, and lowered sex drive. The release of these hormones may provide proper hormonal balance in the brain, which may increase appetite and weight.

Before you can start treatment on this study, you will have "screening tests." These tests will help the study doctor decide if you are eligible to take part in this study. You will have a physical exam, including measurement of your vital signs (blood pressure, heart rate, temperature, and breathing rate). You will be asked to complete 5 questionnaires that will ask about your diagnosis, the medication you are taking, how you have been feeling (such as tense or "wound up"), and any symptoms you may be having (such as pain, poor appetite, weight loss, fatigue, nausea, sleep problems, and depression), and times you have usually gone to bed during the past month. In total, these questionnaires will take about 40 minutes to complete. Women who are able to have children must have a negative urine pregnancy test.

If you are not found to be eligible to take part in this study, you will be provided with a referral to a palliative care doctor who will check your symptoms and plan the appropriate treatment.

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to 1 of 2 groups. You will have an equal chance of being in 1 of the 2 groups. Neither you nor your doctor will know which treatment group you are assigned to. However, in the event of an emergency, for your safety your doctor will be informed about what treatment you are receiving.

Participants in one group will take a specified dose of mirtazapine (with or without food) at bedtime on Days 1-15. On Day 15, you will return to the clinic to repeat the same tests that you had during the screening visit and to be checked for any side effects you may have experienced. You will get 2 more prescriptions (2 different doses--a lesser dose and a greater dose) for mirtazapine. You will then take a lesser dose of mirtazapine (with or without food) for 7 days. During Week 3, you will take the greater dose of mirtazapine for another 7 days until Day 29.

Participants in the other group will take a placebo (a substance that looks like the study drug but has no active ingredients) for 2 weeks. On Day 15, you will return to the clinic to repeat the same tests that you had during the screening visit and to be checked for any side effects you may have experienced. You will be given 2 prescriptions (2 different doses--a lesser dose and a greater dose) for mirtazapine. You will then take a lesser dose of mirtazapine (with or without food) for a 7 days. During Week 3, you will take the greater dose of mirtazapine for another 7 days until Day 29.

You will continue taking part in this study until Day 29, unless the disease gets worse or you experience any intolerable side effects. Otherwise, your participation will end on Day 29, and you will have an end-of-study visit at that time.

Your right arm muscle diameter, your skin fold thickness below your shoulder blade, on the front and back of your right arm, above your right hip bone, and on the front of your right thigh will be measured using a skinfold caliper. The caliper is a device used on the outside of your body to measure skin thickness. You will also be asked to stand on a special scale that will send an extremely low energy, high frequency electrical signal from one foot to your other foot. You will not be able to feel this at all. The device uses the speed at which the signal travels through your body's tissues to calculate body fat weight and body fat percentage. These numbers are used together to determine your body fat, lean body weight, and water content of your body. This will be done on Days 1, 15, and 29.

Participants in both groups will be asked to keep 3 weekly diaries: a food diary, a pill diary recording when mirtazapine is taken, and a daily log of any symptoms that may have been experienced from the cancer before and after treatment began on this study. You will be asked to return to the outpatient clinic at the end of 2 weeks (Day 15) when all tests that were performed during the screening visit will be repeated. All 3 diaries will be reviewed by the research nurse during this clinic visit.

The study nurse will call you on the phone on Days 2 and 16 to find out if you have had increased drowsiness or sleepiness (since the beginning of this study). You will also be called on Days 8 and 22 by the study nurse to check your symptoms, difficulty sleeping, and other side effects you may be experiencing. The phone calls should last about 5-10 minutes each time.

For your end-of-study visit (Day 29), you will return to the outpatient Palliative Care and Rehabilitation Medicine Clinic at M. D. Anderson to be checked on. You will have all of the same tests that you had during the screening visit as well as a review of any side effects you may be experiencing. You will repeat the questionnaires, which should take about 40 minutes to complete. You will need to bring your food diary, pill diary, and symptom log diary to this visit.

All of the study visits will occur on the day listed in this form, or within 3 days earlier or later.

This is an investigational study. Mirtazapine is approved by the FDA (only at the dose levels that will be provided in this study) for depression and commercially available. Its use in this study is experimental. Up to 98 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced cancer patients seen in outpatient clinics or inpatient units at MD Anderson Cancer Center, with presence of anorexia for at least one month, and accompanied by weight loss of > 5 % of pre-illness body weight in the last 6 months. Anorexia on the day of enrollment (day 0 +/-3) must be > 4/10 on ESAS.
2. Patients > 18 years of age
3. Karnofsky Performance score of > 40 at time of inclusion into study
4. Ability to provide informed consent and comply with study procedures
5. Ability and willingness to return to engage in telephone follow-up by research nurse on days 2 (+/- 3 days), 8 (+/- 3 days), 16 ( +/- 3 days), and 22 (+/- 3 days) and return to outpatient clinic for evaluation on days 15 (+/- 3 days), and 29 (+/- 3 days).
6. Negative urine pregnancy test at time of inclusion into study for female patients of childbearing potential, within 24 hours of study enrollment.
7. For patients receiving chemotherapy eligibility to be determined after discussion with primary oncologist
8. Drowsiness of </= 4/10 on ESAS at baseline due to known potential sedating effects of Mirtazapine
9. Patient can continue all medications including complementary therapies or antineoplastic therapy while on-study (with the permission of their Attending MD) if they have been on stable dose for at least 2 weeks.
10. Patients who are on stable doses of antidepressants for at least 2 months.

Exclusion Criteria:

1. Patients who have known dementia or delirium at time of enrollment as determined by a physician.
2. Known hypersensitivity to any ingredient of Mirtazapine
3. Inability to maintain oral intake over the course of the study, such as with mechanical obstruction of the alimentary tract or intractable vomiting
4. Ongoing use of tube feeding or parenteral nutrition
5. Current use of corticosteroids (with the exception of scheduled doses during time of chemotherapy), dronabinol, testosterone and progesterone derivatives such as megestrol acetate, or in the preceding 1 week prior to study enrollment.
6. Pregnancy or lactation or unwillingness to use contraceptives
7. A score of 11 or more, in each subscale of the Hospital Anxiety and Depression scale (HADS) indicating clinical depression or anxiety. Those with HADS scores of > 11 at baseline indicating moderate or severe depression will be excluded from the study and will be referred for appropriate follow up by counselor and psychiatry evaluation.
8. Patients on chronic use of benzodiazepines are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2007-01-08 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of ESAS scores in Appetite | Baseline, and on days (+/-3) 15 and 28
  Primary analysis is a comparison of the difference scores in appetite between baseline and 15 days in the two groups. 2-sample t test used to compare differences between groups or a nonparametric test such as the Wilcoxon test if the data are non-normally distributed. A difference of 2 or more in change scores considered to be clinically meaningful.

SECONDARY OUTCOMES:
Insomnia (as measured by Pittsburgh Sleep Quality Index) | On day 15 ( +/- 3 days), and day 29 ( +/- 3 days)

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Dalal, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Vita G, Compri B, Matcham F, Barbui C, Ostuzzi G. Antidepressants for the treatment of depression in people with cancer. Cochrane Database Syst Rev. 2023 Mar 31;3(3):CD011006. doi: 10.1002/14651858.CD011006.pub4. PMID 36999619
- See also: MD Anderson Cancer Center — http://www.mdanderson.org